CLINICAL TRIAL: NCT05796362
Title: A Randomized, Balanced, Single Dose, Three-treatment, Three-period, Crossover Bioavailability Study of Azithromycin Oleogel in Healthy, Adult, Human Subjects Under Fasting Condition.
Brief Title: A Single-Dose, Three-Way, Three-Sequence, Crossover BA Study of Azithromycin Oleogel
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Principal Investigator, C. Giovanni Traverso MB Bchir PhD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2022p000272
Record Dates: First submitted 2022-09-16; First posted 2023-04-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Infectious Disease; Drug Effect; Clinical Infection
Keywords: Azithromycin; Oleogel; Clinical trial
MeSH Terms: conditions — Communicable Diseases | interventions — Administration, Rectal

STUDY DESIGN:
Intervention Model Description: Randomized, balanced, single dose, three-treatment, three-period, crossover bioavailability study of azithromycin oleogel in healthy, adult, human subjects under fasting condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Reference Azithromycin Tablet (Zithromax) (Active Comparator): 250 mg azithromycin (Zithromax) tablet to be taken once orally.
  Interventions: Drug: Azithromycin Oleogel (Oral and Rectal)
- Oral Oleogel (Experimental): 250 mg azithromycin/ 15 ml oral oleogel (16.67 mg/ml) to be dosed once orally.
  Interventions: Drug: Azithromycin Oleogel (Oral and Rectal)
- Rectal Oleogel (Experimental): 250 mg azithromycin/ 15 ml rectal oleogel (16.67 mg/ml) to be dosed once rectally.
  Interventions: Drug: Azithromycin Oleogel (Oral and Rectal)

INTERVENTIONS:
Drug: Azithromycin Oleogel (Oral and Rectal) — Exploratory study of a novel "oleogel" dosage form of Azithromycin (Zithromax)

SUMMARY:
This is an exploratory study to describe the pharmacokinetics of the azithromycin oral and rectal oleogel in humans compared to the reference oral drug to (Zithromax) assess the impact of the novel formulation on bioavailability. The investigators will perform a randomized, balanced, single dose, three-treatment, three-period, crossover oral bioavailability study under fasted conditions to evaluate the safety and tolerability of azithromycin oleogel and compare the bioavailability of the azithromycin oleogel to the reference drug.

DETAILED DESCRIPTION:
Children have difficulties swallowing tablets including azithromycin (AZT) tablets. In low socioeconomic countries, tablets are typically crushed, dispersed in water, and administered as a suspension to the child. This practice introduces several points of failure, including unpalatability leading to refusal of the drug and lack of clean water for resuspension. Thus, there remains a critical need to develop dosage forms that do not require crushing and suspension. The investigators have developed a formulation inspired by techniques recently described in the field of molecular gastronomy that transform oils into gels, also known as "oleogels". Oils have a prolonged history of use in the food industry, and a very well-established safety profile. Plant-derived oils represent an attractive vehicle for drug delivery. Many drugs have hydrophobic properties and therefore have a greater wettability and solubility in oil in comparison to water. Ingestion of fats stimulates secretion of bile salts and enzymes that enhance drug dissolution in the physiological fluids and drug absorption. Furthermore, converting oils into gels allows for altering the mouth-feel and texture of the dosage form, which affects patient acceptance.

The aim of this exploratory study is to determine azithromycin bioavailability of oral and rectal oleogels in healthy volunteers as well as to make an initial safety evaluation of the oleogels. The reference azithromycin tablet has a bioavailability of 38%, with an AUC of 4.3 mcg*hr/ml, Cmax 0.5 mcg/ml, and Tmax of 2.2 hours. The half-life is approximately 68 hours. The safety profile of azithromycin has been well characterized and single doses of azithromycin are well tolerated, with common reactions including diarrhea/loose stools, nausea, abdominal pain, vomiting, dyspepsia, and vaginitis (all less than 10% of subjects in studies).

The intersubject variability of the pharmacokinetics (PK) parameter estimates for the azithromycin oleogel are derived from our preclinical studies of the azithromycin oleogel in swine; the coefficient of variation for both the oral tablets, oral oleogels, and rectal oleogels are between 30-40%. These estimates of intersubject variability informed our number of subjects, (N=21), for this crossover study. Additional coefficient of variability estimates for oral tablets were found in the literature and were approximately 30%.

Azithromycin is not approved for rectal administration. However, our own studies of the rectal azithromycin oleogel in female Yorkshire swine at doses of 5 mg/kg (40-70 kg weight range) found the following pharmacokinetic parameters: Cmax= 0.224 mcg/ml (CV 35%, n=4); AUC 1.680 mcg*h/ml (CV 30%, n=4). The animals were treated with azithromycin oleogel rectally. After 24 h, tissue mucosal biopsies were collected from the rectum endoscopically under anesthesia. Samples were fixed and stained with Hematoxylin and Eosin and analyzed by a clinical pathologist. Overall, there was no evidence of activity, chronicity, or rectal tissue toxicity in the colorectal mucosa of the rectum in our preclinical swine models, either by gross observation or histologic examination (Table 2). This is in keeping with two exploratory clinical trials of an azithromycin suppository, which did not report any clinically observed or patient-reported safety concerns besides diarrhea at doses of 125-500mg or 1g of azithromycin suppository.

This is an exploratory study to describe the pharmacokinetics of the azithromycin oral and rectal oleogel in humans compared to the reference oral drug to assess the impact of the novel formulation on bioavailability. The investigators will perform a randomized, balanced, single dose, three-treatment, three-period, crossover oral bioavailability study under fasted conditions to evaluate the safety and tolerability of azithromycin oleogel and compare the bioavailability of the azithromycin oleogel to the reference drug. The cross-over design will minimize intersubject variability. Given azithromycin's coefficient of variability, which is estimated to be 30% in humans for the reference drug and 30-60% for the oleogel in swine experiments, the investigators estimate that 21 subjects will be sufficient. This number also accounts for any potential subject dropouts. Due to the half-life of azithromycin being 68 hours, the investigators will give 17 (16-24) days between drug administrations to allow for sufficient wash-out of at least 5 half-lives of azithromycin. Subjects in the study will be closely monitored for any signs of adverse reactions.

Subjects will be given 250mg of azithromycin in each formulation. The maximum recommended dose of azithromycin in humans is 2g in the oral formulation (bioavailability = 38%; effective dose = ~760 mg) or 500mg in the IV formulation. The maximum dose administered to humans is 4g intravenously with the following pharmacokinetic measurements: Cmax 9.91 mcg/ml, AUC 82 mcg*h/ml. At this high dose, side effects seen were most commonly nausea, vomiting, and tinnitus which were mild. In subjects administered 2g intravenous azithromycin, 4 out of 6 developed neutropenia; however, this was not seen at 4g. Based on our non-clinical data in swine with a dosage of 5 mg/kg and a weight range of 40-70 kg, the equivalent human dose would be 4.06-4.89 mg/kg (approximately 305-367 mg for a 75 kg person). The maximum azithromycin a subject would absorb is 250 mg, which is still lower than the 2g dose with 38% bioavailability (~760mg).

Subjects will be screened for up to 28 days prior to first dose. Treatment Period 1 begins with baseline when subjects are admitted to the study center the night before for a 10-hour overnight fast prior to the first dose. After admission, subjects will undergo pre-study evaluations. The subjects will be assigned a subject number before the first study-specific procedure during baseline (e.g., blood sample). A randomization number will be assigned just prior to dosing, after baseline evaluation results have established their continued study eligibility.

After a 10-hour overnight fast, subject will receive a single dose of rectal oleogel test [X] (250mg drug in about 15 ml of oleogel) with continued fast, oral oleogel test [T] (250mg drug in about 15 ml of oleogel), or oral reference tablet [R] with 240 mL of water. For four hours thereafter, subjects should remain in the fasting state and seated in the upright or semi-recumbent position. Brief periods of ambulation are allowed for study-related activities and use of the toilet. Blood samples will be obtained predose and over the next 72 hours. Water will be permitted ad libitum except for one hour before and one hour after dosing. Subjects will be served standardized meals according to a predefined schedule throughout the study.

After approximately a 17-day period away from the study, subjects will return to the study site for Treatment Period 2 and undergo assessments and blood collection similar to Treatment Period 1. The treatment administered will be defined in the randomization schedule.

After approximately a 17-day period away from the study, subjects will return to the study site for Treatment Period 3 and undergo assessments and blood collection similar to Treatment Periods 1 and 2. The treatment administered will be defined in the randomization schedule.

The end-of-study (EOS) evaluation will be performed after completion of the final PK sample following Treatment Period 3 or up to 7 days thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Normal, healthy, adult subjects, 18 to 45 years of age, weight of 45 to 100 kg, and body mass index (BMI) between 18.5 to 30.0 kg/m2.
* Normal hematological, hepatic and renal function as defined by the testing laboratory's normal ranges, and the inclusion of healthy subjects with out-of-range values that fall within a certain range that have no clinical significance for healthy volunteer expansion.
* Willing to use two forms of contraceptive measures or abstinence for the entire duration of the trial.

Exclusion Criteria:

* Participation in an investigational drug or device study within 90 days prior to study drug dosing, i.e., there must be at least 90 days in between the last dose on a prior study and dose administration on this trial.
* Use of tobacco products within the past one year.
* Concomitant disease or condition, including laboratory abnormality, which may interfere with the conduct of the study, or which would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study, including, but not limited to coronary heart disease, diabetes, and adrenal-cortical insufficiency, cancer, alcohol dependency or abuse, drug dependency or abuse, or psychiatric disease.
* Current or past medical condition that might significantly affect the pharmacokinetics of azithromycin.
* Known hypersensitivity to azithromycin, erythromycin, any macrolide or ketolide drug.
* Have history of cholestatic jaundice/hepatic dysfunction associated with prior use of azithromycin.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-08-08 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Azithromycin bioavailability via pharmacokinetics | Up to 10 weeks (17 days on study total)
  Azithromycin bioavailability of oral and rectal oleogels in healthy volunteers as measured by drug concentrations serum of study participants compared to reference standard bioavailability
Initial Azithromycin Oleogel Safety Evaluation | Up to 10 weeks (17 days on study total)
  Initial safety of azithromycin oral and rectal oleogels in healthy volunteers measured by self reported symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No